CLINICAL TRIAL: NCT06457542
Title: Comparative Effects of Active Release Technique and Soft Tissue Mobilization in Shoulder Impingement Syndrome
Brief Title: Comparative Effects of ART and STM in Shoulder Impingement Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Faisalabad (Other)
Collaborators: Allied Hospital Faisalabad (Other)
Responsible Party: Principal Investigator, Fatima Afzaal, Principal investigator, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TUF\DR\SA\MSPP\2024\384
Record Dates: First submitted 2024-05-24; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Shoulder Impingement Syndrome
Keywords: Shoulder impingement syndrome; Active release technique; ROM; Soft tissue mobilization; Pain
MeSH Terms: conditions — Shoulder Impingement Syndrome; Pain

STUDY DESIGN:
Intervention Model Description: Model involves two groups having disease of shoulder impigement syndrome. First group recieves treatment active release technique and Second group recieves soft tissue mobilization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Release Technique (Other): Active release technique is a technique used for to treat impingment syndrome.
  Interventions: Other: Active Release Technique
- Soft Tissue Mobilization (Other): Soft Tissue Moboilization is techniques used for to treat shoulder pain. Soft tissue mobilization (STM) targeting the subscapularis muscle.
  Interventions: Other: Soft Tissue Mobilization

INTERVENTIONS:
Other: Active Release Technique — Active Release Therapy, which involves instructing the patient to sit and then positioning their shoulder in 90-degree abduction. The therapist will provide assistance to the patient's arm and then examine the supraspinous fossa by applying pressure with a finger. The patient will be instructed to gradually bring the arm towards the body as the therapist manipulates the muscle plane. This procedure should be repeated for a duration of 10 minutes, 3 times per week, over a duration of four weeks.
  Arms: Active Release Technique
Other: Soft Tissue Mobilization — Soft Tissue Mobilization (STM) targeting the subscapularis muscle. The participants will be placed in a position where their upper arm bone (humerus) is raised at a 45° angle, with the elbow bent at a 90° angle. Additionally, the humerus will be rotated outward to a position that is normally around 20° to 25° of external rotation. The subscapularis muscle remained examined by touch in the armpit area to locate regions of limited mobility due to myofascial limitations, trigger points or tense bands. The identified limitations remained addressed with STM, which included applying prolonged manual pressure and slow deep stroke to the subscapularis myofascial. This treatment was performed for a period of 7 minutes, three times a week, over a period of four weeks.
  Arms: Soft Tissue Mobilization

SUMMARY:
Shoulder impingement syndrome is primary cause of discomfort and restricted range of motion while reaching above in shoulder region. It is third most common illness affecting musculoskeletal system. The aim of this study will be to analyse comparative effects of active release technique and soft tissue mobilization on pain, range of motion and disability in shoulder impingement syndrome. The study will be a randomized clinical trial. A random sample of 40 subjects with shoulder impingement from Allied hospital, Faisalabad will be evaluated. Subjects who will meet selection criteria will be allocation into two groups by computerized generated allocation method. In addition to ultrasound as baseline treatment group a will receive active release technique while in group B soft tissue mobilization will be administrated for 4 weeks. Treatment session will be 12 session (3 sessions in one week). Baseline, at 2nd week and at 4th week of treatment pain, shoulder elevation, external rotation and shoulder disability will be measure by VAS, goniometer and SPADI. For, data analysis, we will use SPSS software version 23. Data was interrupted through independent t test and repeated measurements ANOVA.

DETAILED DESCRIPTION:
STUDY DESIGN A Randomized Clinical Trial was conducted. SETTING The data of this study was collected from OPD of

* Allied Hospital Faisalabad
* District Headquarter Hospital Faisalabad STUDY DURATION The investigation will be concluded within duration of 4 months subsequent to the acceptance of the synopsis.

STUDY POPULATION Individuals with shoulder impingement syndrome. SAMPLING TECHNIQUE Random Sampling technique

SAMPLE SIZE For size of sample calculation open epi-tool was used by taking overhead reach as main outcome measure (32), and the sample size calculated is 40. These 40 participants were then divided in 2 groups (Group A=20 and group 20). 6 patients will be drop out.

INFORMED CONSENT A signed informed consent from was obtained from the participants before inclusion into the study as it was one of selection criteria. Before obtaining consent all patients in both groups were clearly informed about nature, objectives and duration of study and were assured that their data would not be used for any commercial purpose.

ENROLLENT Availability of signed consent from was considered as the criteria for enrollment to study.

DATA COLLECTION TOOls Visual analogue scale The visual analogue scale will be used to evaluate the level of pain. VAS is dependable besides accurate self-assessment tool that comprises a 10 cm long horizontal line. The scores on this scale range from zero (indicating the absence of pain) to ten (representative the most severe pain possible). The participants were instructed to provide information on the highest level of discomfort they had encountered over the last twenty-four hours. A change of 1.5 points was deemed as the MCID for the Visual Analogue Scale (VAS) The Shoulder Pain and Disability Index (SPADI) is a self-administered survey considered to evaluate the level of pain besides functional impairment caused by shoulder disease. Assessment has a total of thirteen items, divided into two subscales: a pain subscale consisting of five items, and a disability subscale consisting of eight items. The SPADI values ranges from zero to hundred, through a higher number representative a higher level of impairment and disability. Persian iteration of the SPADI questionnaire was used as a dependable and accurate tool, and shown sensitivity to therapeutic modifications in individuals through shoulder ailments. The analysis included the SPADI-pain score, SPADI-disability score, and SPADI-total score. The SPADI total score has been reported to have a MCID ranging from 8 to 13.

Goniometer ROM of the shoulder will be assessed by using a goniometer. The standardized goniometric measures demonstrated excellent consistency within the same rater. The upper limits for shoulder elevation as well as external rotation will be determined.

The patients will be instructed to do maximal range of motion exercises for all arm motions, disregarding any discomfort experienced. The participants will assume a supine position on an examination table during the whole range of movements. Their hips and knees were flexed at an angle of roughly 45°, ensuring that their feet remained level on the table to avoid any curvature of their backs. The elevation was achieved by fully extending the elbow and leading with the thumb. Rotation will be assessed when the shoulder was positioned at a 90° angle of abduction and the elbow was flexed at a 90° angle. Additionally, the forearm will maintain in a neutral position of supination.

SCREENING TESTS Hawkins Kennedy test The Hawkins Kennedy exam will be administered to the patients. The patients will stand with their elbows bent to 90 degrees and their shoulders flexed to 90 degrees, the examiner performs, through passively applying an internally rotation force to arm. A positive result is obtained if the pain is experienced Neer test The sensitivity of this test is 72% and the specificity is 60%. In order to execute the maneuver, the therapist stabilizes the scapula, aligns the arm with the plane of the scapula, and then raises the arm without any active effort from the individual. A positive test result occurs when pain is triggered due to the impingement of the larger tuberosity on the acromion, specifically at an angle between 70 and 110 degrees.

DATA COLLECTION PROCEDURE Subject will screen on basis of inclusion and exclusion criteria. Individuals who have positive screening test and sign consent form will be allocation in to two groups by computerized generated allocation method. Both Group A and B will be given US (Ultrasound) therapy to the subscapularis muscle insertion at the shoulder region, as a baseline treatment. The frequency used is 3 MHz, the intensity used was 0.5 watt/ Cmsq, and the time of the treatment of US was 10 minutes In addition to ultrasound as baseline treatment group a will receive active release technique while in group B soft tissue mobilisation will be administrated for 4 weeks. Treatment session will be 12 session (3 sessions in one week). Baseline, at 2nd week and at 4th week of treatment pain, shoulder elevation, external rotation and shoulder disability will be measure by VAS, goniometer and SPADI.

TREATMENT PLAN Active release technique (ART) Group A will undergo active release therapy, which involves instructing the patient to sit and then positioning their shoulder in 90-degree abduction. The therapist will provide assistance to the patient's arm and then examine the supraspinous fossa by applying pressure with a finger. The patient will be instructed to gradually bring the arm towards the body as the therapist manipulates the muscle plane. This procedure should be repeated for a duration of 10 minutes, 3 times per week, over a duration of four weeks.

Soft tissue mobilization (STM) Group B will receive soft tissue mobilization (STM) targeting the subscapularis muscle. The participants will be placed in a position where their upper arm bone (humerus) is raised at a 45° angle, with the elbow bent at a 90° angle. Additionally, the humerus will be rotated outward to a position that is normally around 20° to 25° of external rotation. The subscapularis muscle remained examined by touch in the armpit area to locate regions of limited mobility due to myofascial limitations, trigger points or tense bands. The identified limitations remained addressed with STM, which included applying prolonged manual pressure and slow deep stroke to the subscapularis myofascial. This treatment was performed for a period of 7 minutes, three times a week, over a period of four weeks SCHEDULE FOR MEASURING OUTCOMES First at baseline then at 2nd week and at 4th week of treatment.

FOLLOW-UPS AND TREATMENT SESSIONS:

Total 12 treatment sessions were done, 3 sessions in one week. STATISTICAL ANALYSIS Using version 23 of SPSS, we will evaluate all of the data. The Shapiro-Wilk test and kurtosis, skewness will be used to evaluate the assumption of data normality. If the data is normally distributed, a parametric test will be used; otherwise, a nonparametric test will be used if the data does not meet the normality assumption.

The current study shows the effects of active release technique (ART) over soft tissue mobilization (STM).The aim of this study was to find out the effects of active realease technique, to find out the effects of soft tissue mobilization and to compare the effects of active release technique and soft tissue mobilization for the patients with shoulder impingment syndrome. This study was a randomized clinical trail (RCT) conducted on a sample convenient sample of 34 shoulder impingment syndrome patients reporting at Allied Hospital Faisalabad from Febuary, 2024 till April, 2024. This study was a Randomized Clinical Trial (RCT) included patients of shoulder impingment syndrome (SIS) selected on the basis on inclusion criteria, patient included into study after filling assessment form that was formed on the basis of inclusion and exclusion criteria, consent was taken from patient and after assessment of patients were randomly allocated into two groups i.e. Group A (Active Release Technique) and Group B (Soft Tissue Moblization). Both groups were followed for the duration of one month, 12 treatment sessions was done. Data collected from the patients were, shoulder pain, ROM of shoulder elevation, external rotation and SPADI questionnaire. Treatment was done to check the effects of interventions for reduction pain and improvement of functional abilities and range of motion of patients of shoulder impingment syndrome, one questionnaire were used for evaluation of pain and functional activities, visual analogue scale for pain, gonimeter for ROM. Primary outcome i.e pain were taken 3 times i.e. at baseline, at 2nd week and after 4th week, while secondary outcome i.e. function and ROM were taken at baseline, at 2nd week and at 4th week. Both treatments are equally effective in decreasing pain and disability. The active release technique and soft tissue mobilization have previously been used for the cure of shoulder pain in clinical settings and in several research studies and always been considered as the best treatment protocol for shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* Age ranges from 40-60 years old
* Unilateral shoulder involvement
* A visual analogue scale (VAS) score of 5 or above
* Abstaining from the use of the painkillers, the anti-inflammatory medicines, and the muscle relaxants for twenty-four hours before to participate
* The Neer test and the Hawkin's test both yielded favorable results
* Every participant volunteered their signature on the informed consent form.

Exclusion Criteria:

* Open wounds at shoulder
* Infection at shoulder site or of shoulder joint,
* Fractures or acute injury
* Current surgeries
* Swelling and rheumatoid arthritis,
* Adhesive capsulitis
* GH joint instability
* Acromioclavicular joint-dysfunction;
* GH joint degenerative joint-disease;
* Cervical radiculopathy;
* Receiving steroid injections
* Receiving of PT intervention for the shoulder discomfort in the previous six months

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-02-17 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Shoulder pain | 7 minutes
  Visual Analogue Scale Minimum Value= 0mm Maximum Value= 10mm

SECONDARY OUTCOMES:
Shoulder range of motion | 10 minutes
  Goniometer Minimum Value= 0 Degree Maximum Value=120 Degree
Shoulder Function | 15 minutes
  Shoulder Pain and Disability Index Minimum Value= 0 Maximum Value= 100

CONTACTS AND LOCATIONS:
Locations (1):
- Fatima Afzaal, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No